CLINICAL TRIAL: NCT01006265
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-finding Study to Evaluate the Efficacy, Safety, and Tolerability of Three Doses of ACT-128800, an Oral S1P1 Receptor Agonist, Administered for Twenty-four Weeks in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Clinical Study to Evaluate the Efficacy, Safety, and Tolerability of ACT-128800 in Patients With Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-058B201
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ACT-128800 Dose 1 (Experimental): ACT-128800 Dose 1
  Interventions: Drug: ACT-128800 Dose 1
- ACT-128800 Dose 2 (Experimental): ACT-128800 Dose 2
  Interventions: Drug: ACT-128800 Dose 2
- ACT-128800 Dose 3 (Experimental): ACT-128800 Dose 3
  Interventions: Drug: ACT-128800 Dose 3
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-128800 Dose 1 — ACT-128800 (Dose 1) administered orally once daily
  Arms: ACT-128800 Dose 1
Drug: Placebo — Matching placebo administered orally once daily
  Arms: Placebo
Drug: ACT-128800 Dose 2 — ACT-128800 (Dose 2) administered orally once daily
  Arms: ACT-128800 Dose 2
Drug: ACT-128800 Dose 3 — ACT-128800 (Dose 3) administered orally once daily
  Arms: ACT-128800 Dose 3

SUMMARY:
This study will assess the efficacy, safety, and tolerability of ACT-128800 in patients with relapsing-remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females
* Diagnosis of RRMS as defined by the revised (2005) McDonald Diagnostic Criteria for Multiple Sclerosis (MS).
* Signed inform consent prior to initiation of any study-mandated procedure.

Exclusion Criteria:

* A diagnosis of MS categorized as primary progressive or secondary progressive or progressive relapsing.
* Patients currently treated for an autoimmune disorder other than MS.
* Contraindications for MRI.
* Ongoing bacterial, viral, or fungal infection.
* History or presence of malignancy.

Additional inclusion and exclusion criteria apply with respect to medical conditions and concomitant treatments which could affect patients' risk from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 464 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2011-06-01 (Actual); Study Completion 2011-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Pharmaceuticals, Study Director — Actelion
Locations (115):
- United States (25):
  - Clinical Investigative Site 3132, Scottsdale, Arizona
  - Clinical Investigative Site 3100, Tucson, Arizona
  - Clinical Investigative Site 3115, Sacramento, California
  - Clinical Investigative Site 3117, Stanford, California
  - Clinical Invesigative Site 3116, Sarasota, Florida
  - Clinical Investigative Site 3101, Indianapolis, Indiana
  - Clinical Investigative Site 3105, Kansas City, Kansas
  - Clinical Investigative Site 3107, Lenexa, Kansas
  - Clinical Investigative Site 3118, Baltimore, Maryland
  - Clinical Investigative Site 3133, Worcester, Massachusetts
  - Clinical Investigator 3136, St Louis, Missouri
  - Clinical Investigative Site # 3135, Newark, New Jersey
  - Clinical Investigative Site 3129, Latham, New York
  - Clinical Investigative Site # 3128, New York, New York
  - Clinical Investigative Site 3127, Schenectady, New York
  - Clinical Investigative Site 3120, Stony Brook, New York
  - Clinical Investigative Site 3119, Raleigh, North Carolina
  - Clinical Investigator 3126, Akron, Ohio
  - Clinical Investigative Site 3113, Cincinnati, Ohio
  - Clinical Investigative Site 3130, Columbus, Ohio
  - Clinical Investigator 3104, Portland, Oregon
  - Clinical Investigative Site 3125, Philadelphia, Pennsylvania
  - Clinical Investigative Site 3112, Burlington, Vermont
  - Clinical Investigative Site 3111, Richmond, Virginia
  - Clinical Investigative Site 3102, Kirkland, Washington
- Australia (2):
  - Clinical Investigative Site # 1001, Fitzroy
  - Clinical Investigative Site 1000, Westmead
- Austria (3):
  - Clinical Investigative Site 1102, Amstetten
  - Clinical Investigative Site 1100, Sankt Pölten
  - Clinical Investigative Site 1101, Vienna
- Belgium (4):
  - Clinical Investigative Site 1201, La Louvière
  - Clinical Investigative Site # 1205, Liège
  - Clinical Investigative Site 1204, Ottignies
  - Clinical Investigative Site 1203, Sijsele-Damme
- Bulgaria (4):
  - Clinical Investigative Site 1302, Sofia
  - Clinical Investigative Site 1301, Sofia
  - Clinical Investigative Site 1303, Varna
  - Clinical Investigative Site 1304, Varna
- Canada (3):
  - Clinical Investigative Site 1401, Burbaby, British Columbia
  - Clinical Investigative Site # 1401, Burnaby
  - Clinical Investigative Site 1400, Ottawa
- Czechia (6):
  - Clinical Investigative Site 1502, Brno
  - Clinical Investigative Site 1506, Jihlava
  - Clinical Investigative Site 1504, Olomouc
  - Clinical Investigative Site 1501, Ostrava-Poruba
  - Clinical Investigative Site 1500, Prague
  - Clinical Investigative Site 1503, Teplice
- Finland (4):
  - Clinical Investigative Site 1600, Helsinki
  - Clinical Investigative Site 1601, Hyvinkää
  - Clinical Investigative Site 1603, Tampere
  - Clinical Investigative Site 1602, Turku
- Clinical Investigative Site 1701, Montpellier, France
- Germany (7):
  - Clinical Investigative Site # 1806, Bayreuth
  - Clinical Investigative 1807, Berlin
  - Clinical Investigative Site 1803, Berlin
  - Clinical Investigative site 1800, Düsseldorf
  - Clinical Investigative Site 1802, Essen
  - Clinical Investigative Site 1805, Homburg/Saar
  - Clinical Investigative Site 1804, Ulm
- Hungary (6):
  - Clinical Investigative Site 1905, Budapest
  - Clinical Investigative Site # 1904, Budapest
  - Clinical Investigative Site 1908, Budapest
  - Clinical Investigative Site 1902, Győr
  - Clinical Investigative Site 1900, Petofi
  - Clinical Investigative Site 1901, Szentpeteri-Kapu
- Israel (4):
  - Clinical Investigative Site 2000, Ashkelon
  - Clinical Investigative Site 2003, Tel Aviv
  - Clinical Investigative Site 2001, Tel Litwinsky
  - Clinical Investigative Site 2002, Ẕerifin
- Italy (6):
  - Clinical Investigative Site 2101, Gallarte
  - Clinical Investigative Site 2104, Genova
  - Clinical Investigative Site # 2106, Milan
  - Clinical Investigative Site 2102, Padua
  - Clinical Investigative Site 2103, Roma
  - Clinical Investigative Site 2105, Siena
- Netherlands (3):
  - Clinical Investigative Site 2203, Breda
  - Clinical Investigative Site 2202, Nijmegen
  - Clinical Investigative Site 2201, Sittard-Geleen
- Poland (4):
  - Clinical Investigative Site 2305, Katowice
  - Clinical Investigative Site 2303, Poznan
  - Clinical Investigative Site 2304, Warsaw
  - Clinical Investigative Site 2302, Wroclaw
- Romania (3):
  - Clinical Investigative Site 2400, Bucharest
  - Clinical Investigative Site 2401, Cluj-Napoca
  - Clinical Investigative Site 2402, Timișoara
- Russia (9):
  - Clinical Investigative Site # 3202, Moscow
  - Clinical Investigative Site # 3203, Nizhny Novgorod
  - Clinical Investigative Site # 3206, Pyatigorsk
  - Clinical Investigative Site # 3204, Saint Petersburg
  - Clinical Investigative Site 3201, Saint Petersburg
  - Clinical Investigative Site 3200, Saint Petersburg
  - Clinical Investigative Site # 3201, Samara
  - Clinical Investigative Site 3209, Saratov
  - Clinical Investigative Site 3208, Ufa
- Serbia (3):
  - Clinical Investigative Site 2501, Belgrade
  - Clinical Investigative Site 2503, Kragujevac
  - Clinical Investigative Site 2502, Niš
- Spain (6):
  - Clinical Investigative Site 2706, Barcelona
  - Clinical Investigative Site 2702, Madrid
  - Clinical Investigative Site 2705, Madrid
  - Clinical Investigative Site 2701, Málaga
  - Clinical Investigative Site 2700, Seville
  - Clinical Investigative Site 2704, Valencia
- Sweden (3):
  - Clinical Investigative Site 2802, Gothenburg
  - Clinical Investigative Site 2800, Stockholm
  - Clinical Investigative Site 2801, Umed
- Switzerland (2):
  - Clinical Investigative Site 2901, Lugano
  - Clinical Investigative Site 2900, Sankt Gallen
- Ukraine (4):
  - Clinical Investigative Site 3302, Chernihiv
  - Clinical Investigative Site 3303, Dnipropetrovsk
  - Clinical Investigative Site 3300, Kyiv
  - Clinical Investigative Site 3304, Odesa
- United Kingdom (3):
  - Clinical Investigative Site 3003, Bristol
  - Clinical Investigative Site 3004, Devon
  - Clinical Investigative Site 3002, London

REFERENCES:
- [Result] Olsson T, Boster A, Fernandez O, Freedman MS, Pozzilli C, Bach D, Berkani O, Mueller MS, Sidorenko T, Radue EW, Melanson M. Oral ponesimod in relapsing-remitting multiple sclerosis: a randomised phase II trial. J Neurol Neurosurg Psychiatry. 2014 Nov;85(11):1198-208. doi: 10.1136/jnnp-2013-307282. Epub 2014 Mar 21. PMID 24659797
- [Derived] Gisleskog PO, Valenzuela B, Scherz T, Burcklen M, Perez-Ruixo JJ, Poggesi I. An Exposure-Response Analysis of the Clinical Efficacy of Ponesimod in a Randomized Phase II Study in Patients with Multiple Sclerosis. Clin Pharmacokinet. 2021 Sep;60(9):1227-1237. doi: 10.1007/s40262-021-01020-2. Epub 2021 Apr 29. PMID 33914286
- See also: A dose-finding study to evaluate the efficacy, safety, and tolerability of three doses of ACT-128800, an oral S1P1 receptor agonist, administered for twenty-four weeks in patients with relapsing-remitting multiple sclerosis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=AC-058B201&attachmentIdentifier=e1d8c0a4-1949-4873-b703-5a8f2bbc4094&fileName=AC-058B201_Additional_result_data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Ponesimod 40 mg: Participants received ponesimod capsules once daily as per up-titration schedule with an initial dose of 10 milligram (mg) ponesimod on Days 1 to 7 followed by first up-titration dose of 20 mg ponesimod on Days 8 to 14 and lastly received 40 mg ponesimod as second up-titration dose on Day 15 to Week 24.
- Ponesimod 20 mg: Participants received ponesimod capsules once daily as per up-titration schedule with an initial dose of 10 mg ponesimod on Days 1 to 7 followed by 20 mg ponesimod on Day 8 to Week 24.
- Ponesimod 10 mg: Participants received ponesimod capsules once daily as per up-titration schedule with a dose of 10 mg ponesimod on Day 1 to Week 24.
- Placebo: Participants received the ponesimod matching placebo tablets once daily for up to Week 24 as per up-titration schedule.
Period: Overall Study
Arm/Group | Ponesimod 40 mg | Ponesimod 20 mg | Ponesimod 10 mg | Placebo
Started | 119 | 116 | 108 | 121
Treated | 119 | 114 | 108 | 121
Completed | 113 | 107 | 99 | 116
Not Completed | 6 | 9 | 9 | 5
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 7 | 5 | 5
Not completed — Administrative reason | 1 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All-randomized analysis set included all randomized participants, whether or not they received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ponesimod 40 mg | Ponesimod 20 mg | Ponesimod 10 mg | Placebo | Total
Number analyzed (Participants) | 119 | 116 | 108 | 121 | 464
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age ( years ) | 36.5 (8.52) | 35.3 (8.52) | 36.9 (9.24) | 36.6 (8.58) | 36.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 79 | 78 | 71 | 85 | 313
  Gender: Male | 40 | 38 | 37 | 36 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 117 | 116 | 108 | 121 | 462
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6 | 12
  White | 114 | 114 | 105 | 114 | 447
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 0 | 1 | 0 | 0 | 1
  Austria | 2 | 2 | 2 | 3 | 9
  Belgium | 2 | 0 | 0 | 0 | 2
  Bulgaria | 5 | 4 | 5 | 5 | 19
  Canada | 3 | 3 | 4 | 3 | 13
  Finland | 6 | 4 | 4 | 6 | 20
  Czech Republic | 14 | 14 | 12 | 12 | 52
  France | 1 | 1 | 1 | 1 | 4
  Germany | 1 | 2 | 1 | 2 | 6
  Hungary | 7 | 7 | 2 | 3 | 19
  Israel | 3 | 2 | 1 | 3 | 9
  Italy | 8 | 7 | 6 | 7 | 28
  Netherlands | 1 | 1 | 2 | 2 | 6
  Poland | 7 | 8 | 10 | 12 | 37
  Romania | 1 | 2 | 3 | 3 | 9
  Russia | 9 | 9 | 8 | 7 | 33
  Spain | 4 | 2 | 3 | 4 | 13
  Serbia | 10 | 10 | 11 | 11 | 42
  Sweden | 5 | 6 | 4 | 6 | 21
  Switzerland | 0 | 2 | 2 | 1 | 5
  United Kingdom | 5 | 5 | 4 | 4 | 18
  Ukraine | 5 | 6 | 5 | 7 | 23
  United States | 20 | 18 | 18 | 19 | 75

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of New T1 Gadolinium-Enhancing (Gd+) Lesions on Magnetic Resonance Imaging (MRI) Scan From Week 12 to Week 24
Description: Cumulative Number of new T1 gadolinium-enhancing (Gd+) lesions per year on magnetic resonance imaging (MRI) scan from Week 12 to Week 24 were reported. Negative binomial (NB) regression analysis on Per protocol analysis set and imputation was applied for the missing data. Here, MS signifies multiple sclerosis.
Time Frame: From Week 12 to 24
Population: Per protocol analysis set included participants of mITT set (randomized participants who received at least one dose of study drug, and had at least one valid post-baseline MRI) who met the criteria for evaluable participants for the analysis of MRI data (participants with Relapsing-remitting multiple sclerosis (RRMS) received study drug until 168 days, two post-baseline MRIs b/w Week 12-24, no forbidden treatment for MS).
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Ponesimod 40 mg | Ponesimod 20 mg | Ponesimod 10 mg | Placebo
Number analyzed (Participants) | 93 | 98 | 88 | 110
Lesions | 1.4 (3.24) | 1.1 (1.96) | 3.5 (7.27) | 6.2 (13.42)
Statistical Analysis 1: Comparison: Ponesimod 40 mg vs Placebo; Test type: Superiority; p < 0.0001, Negative binomial regression model; Treatment effect (rate ratio) = 0.226, 95% CI 2-sided [0.133 to 0.384]
Statistical Analysis 2: Comparison: Ponesimod 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Negative binomial regression model; Treatment effect (rate ratio) = 0.170, 95% CI 2-sided [0.100 to 0.289]
Statistical Analysis 3: Comparison: Ponesimod 10 mg vs Placebo; Test type: Superiority; p = 0.0318, Negative binomial regression model; Treatment effect (rate ratio) = 0.566, 95% CI 2-sided [0.337 to 0.952]

2. Secondary Outcome: Annualized Confirmed Relapse Rate
Description: Relapse: occurrence of acute episode of one or more new symptoms or worsened symptoms of Multiple Sclerosis (MS), not associated with fever/infection and lasting 24 hours after stable 30 days period. Confirmed relapse: increase from baseline at least 0.5 point Expanded Disability Status Scale (EDSS) score or increase of one point in one, two or three Functional Systems (FS), excluding bowel/bladder and cerebral/mental FS. EDSS and FS scores are based on neurological examination for assessing its impairment in MS. Among eight FS, seven are ordinal clinical rating scales ranging from 0-5 or 6 with higher scale indicating overall functional impairment assessing Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel/Bladder and Cerebral functions. Rating individual FS scores is used to rate EDSS with information concerning gait and use of assistance. EDSS is ordinal clinical scale ranges 0 (normal neurological examination) to 10(death due to MS)
Time Frame: Up to 24 weeks
Population: All treated analysis set included all randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Relapse per year
Arm/Group | Ponesimod 40 mg | Ponesimod 20 mg | Ponesimod 10 mg | Placebo
Number analyzed (Participants) | 119 | 114 | 108 | 121
Relapse per year | 0.224 (0.7834) | 0.396 (1.0169) | 0.297 (0.7987) | 0.601 (1.6626)

3. Secondary Outcome: Number of Participants With First Confirmed Relapse as Assessed by Kaplan-Meier Estimate From Baseline to Week 24
Description: Relapse: occurrence of acute episode of one or more new symptoms or worsened symptoms of MS, not associated with fever/infection and lasting 24 hours after stable 30 days period. Confirmed relapse: increase from baseline at least 0.5 point Expanded Disability Status Scale (EDSS) score or increase of one point in one, two or three Functional Systems (FS), excluding bowel/bladder and cerebral/mental FS. EDSS and FS scores are based on neurological examination for assessing its impairment in MS. Among eight FS, seven are ordinal clinical rating scales ranging from 0-5 or 6 with higher scale indicating overall functional impairment assessing Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel/Bladder and Cerebral functions. Rating individual FS scores is used to rate EDSS with information concerning gait and use of assistance. EDSS is ordinal clinical scale ranges 0 (normal neurological examination) to 10(death due to MS). Kaplan-Meier estimate used for Outcome Measure analysis.
Time Frame: Baseline to Week 24
Population: All treated analysis set included all randomized participants who received at least one dose of study drug. Here 'N' (number of participants analyzed) included all participants who were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 40 mg | Ponesimod 20 mg | Ponesimod 10 mg | Placebo
Number analyzed (Participants) | 66 | 71 | 60 | 65
Participants | 10 | 17 | 14 | 25

ADVERSE EVENTS:
Time Frame: Up to 29 weeks (AEs for Treatment duration (24 weeks) and follow up (5 Weeks) on Day 7 and Day 30 after last dose)
Description: All Treated Analysis set included all randomized participants who received at least one dose of study drug.
Arm/Group | Ponesimod 40 mg | Ponesimod 20 mg | Ponesimod 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/114 | 0/108 | 0/121
Serious Adverse Events (participants affected / at risk) | 3/119 | 7/114 | 7/108 | 5/121
Other Adverse Events (participants affected / at risk) | 83/119 | 73/114 | 69/108 | 77/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ponesimod 40 mg (N=119) | Ponesimod 20 mg (N=114) | Ponesimod 10 mg (N=108) | Placebo (N=121)
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1 | 2 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Macular Oedema (Eye disorders) | 0 | 2 | 0 | 0
Papilloedema (Eye disorders) | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Anaphylactoid Reaction (Immune system disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Measles (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 1 | 0
Nuclear Magnetic Resonance Imaging Abnormal (Investigations) | 0 | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ponesimod 40 mg (N=119) | Ponesimod 20 mg (N=114) | Ponesimod 10 mg (N=108) | Placebo (N=121)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 5 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 1 | 3 | 3
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 3
Eye Pain (Eye disorders) | 0 | 0 | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3 | 8
Dry Mouth (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 6
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3 | 0
Asthenia (General disorders) | 3 | 1 | 1 | 4
Chest Discomfort (General disorders) | 4 | 5 | 0 | 3
Disease Progression (General disorders) | 11 | 9 | 10 | 6
Fatigue (General disorders) | 6 | 9 | 7 | 7
Oedema Peripheral (General disorders) | 13 | 3 | 2 | 2
Pain (General disorders) | 0 | 0 | 0 | 3
Bronchitis (Infections and infestations) | 5 | 4 | 4 | 3
Gastroenteritis (Infections and infestations) | 1 | 3 | 5 | 4
Influenza (Infections and infestations) | 5 | 3 | 3 | 2
Nasopharyngitis (Infections and infestations) | 13 | 12 | 16 | 17
Oral Herpes (Infections and infestations) | 2 | 0 | 2 | 6
Rhinitis (Infections and infestations) | 0 | 4 | 3 | 1
Sinusitis (Infections and infestations) | 6 | 5 | 4 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 9 | 4 | 11
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 2 | 6
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 0
Alanine Aminotransferase Increased (Investigations) | 7 | 7 | 4 | 1
Blood Cholesterol Increased (Investigations) | 2 | 3 | 3 | 1
Forced Expiratory Volume Decreased (Investigations) | 3 | 2 | 2 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 3 | 0
Pulmonary Function Test Decreased (Investigations) | 5 | 0 | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 2 | 6
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 5
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 1
Dizziness (Nervous system disorders) | 11 | 7 | 8 | 3
Headache (Nervous system disorders) | 15 | 16 | 15 | 18
Hypoaesthesia (Nervous system disorders) | 3 | 2 | 2 | 2
Migraine (Nervous system disorders) | 5 | 3 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 3 | 1
Affect Lability (Psychiatric disorders) | 0 | 0 | 0 | 3
Anxiety (Psychiatric disorders) | 4 | 3 | 5 | 0
Depression (Psychiatric disorders) | 4 | 3 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 4 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 7 | 5 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 4 | 4

LIMITATIONS AND CAVEATS:
No limitation was identified for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.